CLINICAL TRIAL: NCT06328179
Title: Clinical Study Protocol for the Treatment of Newly Diagnosed and Relapsed/Refractory Acute Myeloid Leukemia With KMT2A Gene Abnormalities Using VHEA（Venetoclax With Homoharringtonine，Etoposide，Cytarabine）
Brief Title: Clinical Study Protocol for the Treatment of ND-AML and RR-AML With KMT2A Gene Abnormalities Using VHEA.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huai'an First People's Hospital (Other)
Collaborators: Zhenjiang First People's Hospital (Other); The First People's Hospital of Changzhou (Other); The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY-2023-058-01
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Cytarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VHEA regimen in the treatment of ND-AML and RR-AML with MLL gene abnormalities. (Experimental): Venetoclax 100 mg d1，200 mg d2，400 mg d3-14； homoharringtoine, HHT 2 mg/m2，qd，d1-7； Etoposide 0.1 g，qd，d1-5； Cytarabine 100 mg/m2，qd，d1-7
  The patient meets the criteria for autologous hematopoietic stem cell transplantation (ASCT) during the treatment process, they can undergo ASCT.If the patient meets the criteria for transplantation and there is a suitable donor, they can undergo allogeneic hematopoietic stem cell transplantation (allo-HSCT).
  Interventions: Drug: Venetoclax 100 mg d1，200 mg d2，400 mg d3-14；

INTERVENTIONS:
Drug: Venetoclax 100 mg d1，200 mg d2，400 mg d3-14； — VHEA -Induction Phase Regimen/Consolidation therapy after remission
  Other Names: Homoharringtoine, HHT 2 mg/m2，qd，d1-7; Etoposide 0.1 g，qd，d1-5; Cytarabine 100 mg/m2，qd，d1-7

SUMMARY:
This study is a clinical trial aimed at evaluating the efficacy and safety of the VHEA（Venetoclax with Homoharringtonine，Etoposide，Cytarabine）regimen in the treatment of newly diagnosed and relapsed/refractory acute myeloid leukemia (AML) with MLL gene abnormalities.

This study includes the induction and consolidation phases of AML treatment.

DETAILED DESCRIPTION:
This study is a multicenter, single-arm, open-label clinical trial aimed at evaluating the efficacy and safety of the VHEA（Venetoclax with Homoharringtonine，Etoposide，Cytarabine）regimen in the treatment of newly diagnosed and relapsed/refractory acute myeloid leukemia (AML) with MLL gene abnormalities.

Leukemia is a malignant tumor of the blood system that seriously endangers human health, ranking among the top 10 in the mortality rate of malignant tumors in all age groups in China. Acute myeloid leukemia (AML) is a malignant clonal blood system disease originating from hematopoietic stem and progenitor cells, accounting for about 35% of newly diagnosed leukemia cases each year and 80% of adult leukemia cases. The overall prognosis is poor, with approximately 10-40% of newly diagnosed AML patients unable to achieve CR, and over 50% of AML patients eventually relapse. Especially in AML with KMT2A gene abnormalities, the conventional "3+7" chemotherapy regimen has a low remission rate and a high relapse rate.

Chromosomal translocations include the Mixed Lineage Leukemia gene (MLL), also known as the KMT2A gene, which produces various MLL fusion genes, including AF4, AF6, AF9, AF10, ENL, ELL, and AF1q. Currently, more than 70 MLL fusion genes have been reported. MLL gene abnormalities associated with leukemia account for 5% to 10% of all acute leukemias, and MLL-related leukemia has a poor prognosis. There is currently no standard treatment regimen for MLL-related AML with good efficacy. Current treatment options include conventional chemotherapy, targeted epigenetic and DNA damage response therapies. Conventional chemotherapy includes regimens composed of anthracyclines, cytarabine, and etoposide, followed by consolidation therapy with allogeneic hematopoietic stem cell transplantation, but the efficacy is still unsatisfactory.

Based on preliminary data from our institution, there have been a total of 30 cases of AML with MLL gene abnormalities since 2016, accounting for approximately 12% of all AML cases. Among these, 14 cases received initial induction chemotherapy using the standard "3+7" regimen, with only 4 cases achieving complete remission (28.6%), 3 cases achieving partial remission (21.4%), and 7 cases showing no response (50%). Five cases received induction chemotherapy using a priming regimen, but none achieved remission. Additionally, 11 patients either refused chemotherapy or sought treatment at other hospitals, indicating that conventional chemotherapy regimens do not yield satisfactory results in AML patients with MLL gene abnormalities. Therefore, it is of great clinical significance to explore more effective chemotherapy regimens for MLL gene abnormality-associated acute leukemia.

Venetoclax has demonstrated anti-tumor activity in various hematologic malignancies. In November 2018, the U.S. Food and Drug Administration (FDA) approved the use of Venetoclax in combination with hypomethylating agents (HMAs) or low-dose cytarabine for newly diagnosed AML patients aged 75 years and older who are unfit for intensive chemotherapy. According to the 2021 NCCN guidelines, Venetoclax in combination with HMAs or low-dose cytarabine is an important treatment strategy for both newly diagnosed elderly AML patients and relapsed/refractory AML patients who are not suitable for intensive chemotherapy. Recent exploratory studies have also been conducted on the use of Venetoclax in combination with hypomethylating therapy in newly diagnosed and relapsed/refractory AML with KMT2A gene rearrangement. These studies found that Venetoclax in combination with decitabine or azacitidine achieved an overall response rate (ORR) of 83% and a complete response/complete response with incomplete hematologic recovery (CR/CRi) of 75% in newly diagnosed AML with KMT2A gene rearrangement. However, in relapsed/refractory AML with KMT2A rearrangement, the ORR and CR/CRi were only 17% and 8%, respectively.

Homoharringtonine (HHT) is widely used for the treatment of myeloid leukemia. HHT promotes apoptosis and inhibits autophagy in CML cells by activating ERK phosphorylation and inhibiting Akt phosphorylation. Bcl-2 protein is an apoptosis inhibitor that plays an important regulatory role in cell apoptosis. NFκB is a nuclear transcription factor present in cells that regulates κ immunoglobulin and has anti-apoptotic effects. HHT significantly inhibits the expression of NFκB and Bcl-2 protein, ultimately leading to cell apoptosis.

Venetoclax has been widely used in various hematological malignancies, but the short duration of sustained remission and the occurrence of resistance are the main problems currently. The mechanisms of Venetoclax resistance mainly include the activation of selective dependence on the Bcl-2 anti-apoptotic protein family and kinase mutations, among which other members of the Bcl-2 family, including BCL2-A1, MCL-1, and BCL-XL, have been proven to be key factors leading to primary or acquired resistance to Venetoclax. Recent studies have shown that Venetoclax has synergistic inhibition of AML cell proliferation with Homoharringtonine, reduces mitochondrial membrane potential, promotes AML cell apoptosis, and exhibits time-dependent and concentration-dependent effects. Venetoclax with Homoharringtonine can synergistically promote apoptosis of AML cell lines and primary cells by inhibiting the activation of the MAPK/ERK, PI3K/AKT, and P53 signaling pathways. Therefore, based on this, we propose that Venetoclax with Homoharringtonine, Etoposide, and Cytarabine may be an effective treatment option for newly diagnosed and relapsed/refractory AML with MLL gene abnormalities.

This study will include AML patients with newly diagnosed or relapsed refractory MALL gene abnormalities. The VHEA regimen will be used for induction, followed by one consolidation cycle after achieving CRh/CRi/MLFS. If patients have a PR/NR, VHEA will be continued for induction therapy until disease remission. After achieving remission, patients who are willing and meet the criteria will undergo transplantation. If transplantation is not performed, consolidation chemotherapy will be continued until disease progression.

Specific treatment plan: VHEA Venetoclax 100 mg d1，200 mg d2，400 mg d3-14； homoharringtoine, HHT 2 mg/m2，qd，d1-7； Etoposide 0.1 g，qd，d1-5； Cytarabine 100 mg/m2，qd，d1-7

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years old;Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Expected survival time of at least 3 months.
* Does not meet any of the following criteria for severe heart, lung, liver, or kidney disease:A) History of congestive heart failure requiring treatment, or ejection fraction ≤ 50%, or presence of chronic stable angina;B) Lung diffusing capacity for carbon monoxide (DLCO) ≤ 65%, or forced expiratory volume in one second (FEV1) ≤ 65%;C) Moderate liver dysfunction, total bilirubin > 1.5 to ≤ 3.0 × upper limit of normal (ULN);D) Creatinine clearance ≥ 30 mL/min to < 45 mL/min.
* No other significant contraindications to chemotherapy as determined by the physician;
* Capable of understanding and willing to sign the informed consent form for this study.

Exclusion Criteria:

* Presence of other malignancies;
* Underwent cardiac vascular intervention or stent placement within 12 months prior to signing the informed consent, or history of myocardial infarction, unstable angina, or other clinically significant cardiac disease;
* Uncontrolled active infection (including bacterial, fungal, or viral infection) and visceral bleeding;
* Pregnant or lactating women;
* Participation in any other clinical study within 3 months prior to signing the informed consent;
* Any other condition deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate，ORR | The period of 1 year from the start of treatment.
  The morphological efficacy evaluation of the subjects is divided into four outcomes: complete remission (CR), complete remission with partial hematologic recovery (CRh), complete remission with incomplete hematologic recovery (CRi), partial remission (PR), and no remission (NR). Among them, CR, CRh, CRi, MLFS, and PR are collectively referred to as ORR. The evaluation time point is on the 21st day after the start of chemotherapy. When the patient is first evaluated as CR/CRh/CRi, complete test results such as peripheral blood, bone marrow, and clinical symptoms are required.

SECONDARY OUTCOMES:
Overall survival, OS | The period of 1 year from the start of treatment.
  The evaluation of overall survival (OS) is measured from the date of the first VHEA regimen until the date of death from any cause. For subjects who are still alive at the last follow-up, their OS is censored at the time of the last follow-up. For subjects lost to follow-up, their OS is censored at the last confirmed alive time before the loss to follow-up.
Event free survival, EFS | The period of 1 year from the start of treatment.
  The evaluation of event-free survival (EFS) is measured from the date of the first VHEA regimen to the date of treatment failure, disease relapse, or death for any reason. For subjects who are still alive at the last follow-up, their EFS is considered as censored at the last follow-up time. For subjects lost to follow-up, their EFS is considered as censored at the last confirmed alive time before the loss to follow-up.
Duration of remission, DOR | The period of 2 year from the start of treatment.
  Duration of response (DoR) is the time from the initial achievement of complete.

OTHER OUTCOMES:
Adverse event, AE | The period of 1 year from the start of treatment.
  Evaluate the incidence and severity of grade 3-4 adverse events (AE) in the VHEA
Treatment-related mortality, TRM | The period of 1 year from the start of treatment.
  This includes any deaths caused by any reason, including deaths related to disease treatment in a complete response (CR) state or deaths occurring within 28 days of starting treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Huaian No.1 People's Hospital of Nanjing Medical University（Huai'an First People's Hospital）, Huai'an, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided